CLINICAL TRIAL: NCT03726255
Title: Retrospective Evaluation of Stem Cell Therapy: a Compassionate Use Program in Perianal Fistula.
Brief Title: Stem Cell Therapy: a Compassionate Use Program in Perianal Fistula
Acronym: RESCeCUF
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Other Study IDs: EO166-18_FJD
Record Dates: First submitted 2018-10-26; First posted 2018-10-31 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-10

CONDITIONS: Perianal Fistula
Keywords: Perianal fistula; compassionate use; mesenchymal stem cells

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stromal Vascular fraction: 31 patients were treated with one injection of Stromal Vascular Fraction from adipose tissue obtained by liposuction. Procedure: curettage, closure of the internal opening (IO) and SVF injection in IO (50%) and fistula tract (50%)
  Interventions: Procedure: Mesenchymal Stem Cell injection
- Autologous mesenchymal stem cells: 9 patients were treated with one injection of autologous mesenchymal stem cells from adipose tissue. Procedure: curettage, closure of the internal opening (IO) and autologous cell injection in IO (50%) and fistula tract (50%)
  Interventions: Procedure: Mesenchymal Stem Cell injection
- Allogenic mesenchymal stem cells: 12 patients were treated with one injection of allogenic mesenchymal stem cells of healthy donors: Procedure: curettage, closure of the internal opening (IO) and allogenic cell injection in IO (50%) and fistula tract (50%)
  Interventions: Procedure: Mesenchymal Stem Cell injection

INTERVENTIONS:
Procedure: Mesenchymal Stem Cell injection — curettage, closure of the internal opening (IO) and cell injection in IO (50%) and fistula tract (50%)

SUMMARY:
This observational study aims at assessing the safety and efficacy profiles of mesenchymal stem cell, in different formats (SVF, autologous, allogenic), to treat complex perianal fistula according to the Spanish national Compassionate-use law .

DETAILED DESCRIPTION:
Under controlled circumstances, and approved by European and Spanish laws, a Compassionate-use Program allows the use of stem-cell therapy for patients with non-healing diseases, mostly complex fistula-in-ano, who do not meet criteria to be included in a clinical trial. Candidates had previously undergone multiple surgical interventions that had failed. The intervention consisted of surgery (with closure of the internal opening or a surgical flap performance), followed by stem cells injection. Three types of cells were used for implant: stromal vascular fraction, autologous expanded adipose-derived or allogenic adipose derived stem cells.

Healing was evaluated at 6th month follow-up. Outcome was classified as partial response or healing. Relapse was evaluated 1 year later. Maximum follow up period was 48 months.

ELIGIBILITY:
Inclusion Criteria:

* patients with complex perianal fistula
* patients who didn't meet criteria of the clinical trial (CT) in development
* foreign patients, who were not allowed to be included in the CT
* patients included in some CT control arms
* failure treatment in patients included in a CT treatment arm as a retreatment

Exclusion Criteria:

* not signature informed consent

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We present an observational study, including 52 cases (53% male and 47% female) treated by a compassionate use ASC program. The mean age was 45 years and ranged from 24 to 69 years. There were 42 perianal fistulas, 7 rectovaginal fistulas, 1 urethrorectal fistula, 1 sacral fistula and 1 hidradenitis suppurativa. All the cases had previous failed surgeries. Thirteen of fifty-two (25%) of the cases presented fecal incontinence at the moment of enrollment. 5/52 (9,6%) of the cases presented anal stenosis and 11/52 (21%) had a scaring anus.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Number of patients with fistula healed | 12 months
  Complete closure of the fistula and epithelization of the external orifice

SECONDARY OUTCOMES:
Number of adversus events | 12 months
  general adversus events

CONTACTS AND LOCATIONS:
Overall Officials: Damian Garcia-Olmo, Prof., Principal Investigator — Instituto de Investigación Sanitaria Fundación Jiménez Díaz
Locations (1):
- Instituto Investigación Sanitario Fundación Jiménez Díaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No